CLINICAL TRIAL: NCT00761254
Title: Oral Domperidone for Relief of Gastrointestinal Disorders in Patients Who Failed Standard Therapy
Brief Title: Domperidone for Relief of Gastrointestinal Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI withdrew due to increased responsibilities in clinical department.
Sponsor: Carle Physician Group (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-153
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Gastroparesis; GERD; Esophagitis; Dyspepsia; Chronic Idiopathic Constipation; Nausea; Vomiting
Keywords: Domperidone; Gastroparesis
MeSH Terms: conditions — Gastroparesis; Gastroesophageal Reflux; Esophagitis; Dyspepsia; Nausea; Vomiting | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Domperidone — Initially, 10mg of oral Domperidone will be administered 2-4 times a day as needed. This dosage may be increased or decreased depending on how the subject responds to the drug.
  Other Names: Motilium

SUMMARY:
The purpose of this study is to make Domperidone available to patients with gastrointestinal disorders who have failed standard therapy and who might benefit from it.

DETAILED DESCRIPTION:
Domperidone is the only medication that is a true prokinetic with a low percentage of side effects that is useful in the treatment of certain GI conditions, including gastroparesis and other motility disorders.

According to recent regulations, writing prescriptions for subject to obtain domperidone outside the United States has been determined to be illegal and the FDA has issued warnings against pharmacies compounding domperidone. The legal way of administering domperidone is by obtaining an Investigational New Drug Application.

This study is an effort to both follow federal regulations and provide the medication to subjects who would benefit from it where standard therapy has failed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* symptoms or manifestations secondary to GERD (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms, gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that is refractory to standard therapy
* subjects must have a comprehensive evaluation to eliminate other causes of their symptoms.

Exclusion Criteria:

* history of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation, and Torsade de pointes. Subjects with minor forms of ectopy (PACs) are not necessarily excluded.
* clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTc > 450 milliseconds for males, QTc > 470 milliseconds for females.)
* clinically significant electrolyte disorders.
* gastrointestinal hemorrhage or obstruction.
* presence of a prolactinoma (prolactin-releasing pituitary tumor.)
* pregnant or breast feeding female.
* known allergy to Domperidone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Relief for patients with gastrointestinal disorders who have failed standard therapy | As long as the subjects continue to take Domperidone.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Batey, M.D., Principal Investigator — Carle Health Care Incorporated d/b/a Carle Physician Group; Anna Keck, PhD, Study Director — Carle Foundation Hospital; James Dougherty, MD, Study Director — Carle Foundation Hospital; Eugene Greenberg, MD, Principal Investigator — Carle Physician Group; Vicki Shah, PA, Principal Investigator — Carle Physician Group
Locations (1):
- Carle Health Care Incorporated d/b/a Carle Physician Group, Urbana, Illinois, United States

REFERENCES:
- [Background] Ahmad N, Keith-Ferris J, Gooden E, Abell T. Making a case for domperidone in the treatment of gastrointestinal motility disorders. Curr Opin Pharmacol. 2006 Dec;6(6):571-6. doi: 10.1016/j.coph.2006.07.004. Epub 2006 Sep 25. PMID 16997628
- [Background] Reddymasu SC, Soykan I, McCallum RW. Domperidone: review of pharmacology and clinical applications in gastroenterology. Am J Gastroenterol. 2007 Sep;102(9):2036-45. doi: 10.1111/j.1572-0241.2007.01255.x. Epub 2007 May 3. PMID 17488253
- [Background] Barone JA. Domperidone: a peripherally acting dopamine2-receptor antagonist. Ann Pharmacother. 1999 Apr;33(4):429-40. doi: 10.1345/aph.18003. PMID 10332535
- [Background] Champion MC, Hartnett M, Yen M. Domperidone, a new dopamine antagonist. CMAJ. 1986 Sep 1;135(5):457-61. PMID 3527396